CLINICAL TRIAL: NCT04412850
Title: Role of Intravenous Magnesium Sulphate in Improving Clinical Outcome in Patients Suffering From Acute Ischemic Stroke
Brief Title: Intravenous Magnesium Sulphate in Acute Ischemic Stroke
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Huda Naim, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: huda01
Record Dates: First submitted 2020-05-11; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Stroke; Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Experimental): Magnesium will be given intravenously with a loading dose of 4 g in 50 mL saline over a 15-minute period and 16 g in 100 mL over a 24-hour period in a continuous-infusion form. The regiment chosen for this study is designed to double serum magnesium concentration to twice physiological concentration for therapeutic effects in humans, Serum levels between 4.8mg/dl-6mg/dl are considered to have an optimal neuroprotective effect.
  Interventions: Drug: Magnesium Sulfate
- placebo group (Placebo Comparator): Normal Saline in equal volume as the control group.
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — Magnesium and placebo (Normal Saline) will be prepared as solutions of identical volume and appearance. All patients will be randomized and blind to treatment.
  All patients will have pretreatment Electrogram (ECG), serum biochemistry and serum Magnesium levels. Serum Magnesium levels will also be measured at 48 hours. Blood pressure, heart rate, respiratory rate and serious adverse events will be monitored at baseline, 15 minutes, and 12, 24 and 48 hours after infusion. Magnesium will be given intravenously with a loading dose of 4 g in 50 mL saline over a 15-minute period and 16 g in 100 mL over a 24-hour period in a continuous-infusion form.
  Follow-up visits will be conducted by the same investigators, and repeated scores on the NIH Stroke Scale will be obtained at 24 hours, 48 hours post admission and on the day of discharge.

SUMMARY:
Magnesium has a neuroprotective role so the investigators aim to evaluate the role of intravenous magnesium sulphate in improving the clinical outcomes as assessed by the NIH Stroke Scale (NIHSS) in patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a confirmed diagnosis of ischemic stroke on neurological examination and CT scan findings aged between 45 -95 years of age of either gender.
* Adults presenting within a stroke onset of 24 hours.

Exclusion Criteria:

* Patients with confirmed diagnosis other than ischemic stroke (evidence of Intracranial bleed or space occupying lesion)

  * Subjects with systolic blood pressure less than 90mmHg
  * Presence of Bundle Branch block or atrioventricular block.
  * Serum Creatinine > 3mg/dl
  * Respiratory failure (O2 saturation <90% or Respiratory Rate >24 or <12)
  * Pregnancy.

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Improvement In Clinical Outcome As Measured By The improvement in NIH Stroke Scale After Infusion Of Magnesium Sulphate In Patients Suffering From Acute Ischemic Stroke. | 7 days

SECONDARY OUTCOMES:
adverse effects | 7 days

IPD SHARING:
Plan to Share IPD: No